CLINICAL TRIAL: NCT06743828
Title: Impacts of Fermented Pea- and Legume-based Product High in Protein on Gut Microbiota and Health: a Randomized, Single-blinded, Controlled, Cross-over Trial
Brief Title: Impacts of Fermented Pea- and Legume-based Product on Gut Microbiota and Health
Acronym: HealthFerm
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: University of Turku (Other); Umeå University (Other); KU Leuven (Other); Flemish institute of biotechnology (VIB) (Other); ETH Zurich (Other)
Responsible Party: Principal Investigator, Marjukka Kolehmainen, Professor, University of Eastern Finland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 159/2024 HealthFerm
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Syndrome
Keywords: Fermentation; Plant Proteins, Dietary; Inflammation Mediators; Gastrointestinal Microbiome; Tryptophan; Cardiometabolic Health
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fermented product (Experimental): Participants consume a fermented pea- and legume-based product daily for three weeks within their diet.
  Interventions: Other: Fermented meat alternative
- Unfermented product (Active Comparator): Participants consume an unfermented pea- and legume-based product daily for three weeks within their diet.
  Interventions: Other: Unfermented meat alternative
- Habitual diet (No Intervention): Participants consume their habitual diet without any intervention products.

INTERVENTIONS:
Other: Fermented meat alternative — Participants incorporate a novel fermented product into their habitual diet for three weeks. The product replaces the main protein source of the meal(s). Participants will receive dietary guidance on how to follow the intervention diet, as well as potential supplement recommendations provided by the authorized nutritionist.
  Arms: Fermented product
Other: Unfermented meat alternative — Participants incorporate an unfermented product into their habitual diet for three weeks. The product replaces the main protein source of the meal(s). Participants will receive dietary guidance on how to follow the intervention diet, as well as potential supplement recommendations provided by the authorized nutritionist.
  Arms: Unfermented product

SUMMARY:
This study aims to investigate the effects of consuming fermented pea- and legume-based product on gut and overall human health. It is a randomized, single-blinded, controlled, cross-over trial with a dietary intervention.

A total of 100 participants will be enrolled in this study and they will eat both fermented and unfermented pea- and legume-based products for three weeks. Participants will eat their habitual diet between the dietary intervention periods (wash-out).

During the study, participants' perceived health, inflammatory markers, glucose and lipid metabolism, tryptophan metabolites, gastrointestinal symptoms, and gut microbiota will be assessed.

DETAILED DESCRIPTION:
Plant-based protein sources, such as those derived from peas and legumes, are experiencing high demand due to their role in reducing reliance on animal products and promoting a more sustainable food system. Despite this, there is limited information available regarding the impact of components like fibre in plant-based foods on protein and other nutrients' metabolism. In addition, the evidence of the health effects of meat alternatives is still scarce.

Food fermentation emerges as a potential solution to enhance the absorption of plant-based protein and various nutrients in the small intestine. This is achieved by reducing antinutrients and facilitating the absorption process. Additionally, food fermentation has implications for the composition and metabolic activity of the gut microbiota, influencing metabolism, immune responses, intestinal function, and overall health. The metabolism of tryptophan in the gut, modulated by the gut microbiota and the production of various metabolites, may serve as a key link in these observed health effects.

The fermentation of plant-based foods potentially enhances their beneficial health effects, and investigating this contributes to an increased understanding of the gut-mediated health effects of foods and the mechanisms behind them. This study is part of a European research project HealthFerm.

Detailed objectives are to:

1. compare fermented and unfermented pea- and legume-based food products on blood lipid and glucose metabolism and gastrointestinal comfort as well as perceived and observed overall well-being.
2. study the effects of fermented and unfermented pea- and legume-based food consumption on gut permeability and inflammation markers.
3. study the difference in microbiota composition, diversity, and its contribution to cardiometabolic outcomes after consuming fermented and unfermented pea- and legume-based food products .
4. study the difference in microbiota-related metabolites, especially tryptophan metabolites, between fermented and unfermented pea- and legume-based food products.

A total of 100 participants will be enrolled in this randomized, single-blinded, controlled, cross-over trial, during which they will eat both fermented and unfermented pea- and legume-based products as part of their habitual diet. The study follows this sequence:

Weeks 1-3: Habitual diet Weeks 4-6: Intervention diet 1 Weeks 7-9: Habitual diet (wash-out) Weeks 10-12: Intervention diet 2

Fasting blood, urinary and faecal samples, as well as food diaries and questionnaires, are collected at the end of each study period to assess participants' diet, perceived health, gastrointestinal symptoms, inflammatory markers, glucose and lipid metabolism, tryptophan metabolites, and gut microbiota composition and their metabolites, such as short-chain fatty acids. In addition, participants' values and attitudes towards fermented foods are assessed. At the end of the study, participants will receive their laboratory results and dietary guidance for their habitual diet from a registered dietitian.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference >90 cm (women) or >100 cm (men) OR BMI 27-35 kg/m2
* One of the following:

  * raised blood pressure (systolic ≥ 130 mmHg and/or diastolic 85 mmHg)
  * raised fasting plasma glucose (≥ 5.6 mmol/l)
  * raised triglycerides (≥ 1.7 mmol/l)
  * raised total cholesterol (≥ 5 mmol/l)
  * raised LDL (≥ 3 mmol/l)
  * reduced HDL (women < 1.3 mmol/l, men 1.0 mmol/l)
* Consumption of at least one meal where the main protein source is meat, fish, or meat alternative on most days
* Willingness to follow intervention diets for the whole study

Exclusion Criteria:

* Diagnosed chronic diseases and conditions which could hamper the adherence to the dietary intervention protocol, e.g., type 1 or 2 diabetes, chronic liver, thyroid, kidney, or gastrointestinal diseases
* Pregnancy and lactation
* Gluten-free or vegan diet
* Recent use of antibiotics (within 3 months)
* Gastrointestinal surgery (within 6 months)
* Alcohol abuse (AUDIT ≥ 15 p and measures of liver function)
* regular smoking or use of snus or nicotine bags

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
P-hs-CRP (mg/l) | Weeks 3, 6, 9, and 12
IL-22 | Weeks 3, 6, 9, and 12
LBP (μg/ml) | Weeks 3, 6, 9, and 12

SECONDARY OUTCOMES:
Changes in the composition gut microbiota | Weeks 3, 6, and 12
  Composition of gut microbiota will be analysed from faecal samples
Short-chain fatty acids assessed from plasma samples | Weeks 3, 6, 9, and 12
Glucose metabolism | Weeks 3, 6, 9, and 12
  fP-Gluk and B-HbA1C (mmol/l)
fP-Insu (mU/l) | Weeks 3, 6, 9, and 12
Lipid metabolism | Weeks 3, 6, 9, and 12
  fP-Kol, fP-Kol-HDL, fP-Kol-LDL, fP-Trigly, and fP-FFA (mmol/l)
Tryptophan metabolism | Weeks 3, 6, 9, and 12
  Tryptophan metabolites will be analysed with non-targeted metabolomics.
Self-reported overall health (Short Form-36 Health Survey, SF-36) | Weeks 3, 6, 9, and 12
  Different sections are rated from 0 to 100 points, where higher scores mean better perceived health.
Self-reported mental health (General Health Questionnaire-12, GHQ-12) | Weeks 3, 6, 9, and 12
  The questionnaire is rated from 0 to 12 points, where higher score means greater psychological distress.
Self-reported gastrointestinal symptoms (Gastrointestinal Symptoms Rating Scale, GSRS) | Weeks 3, 6, 9, and 12
  Different symptoms in the questionnaire are rated from 0 to 7, where higher score means greater symptoms.

OTHER OUTCOMES:
Attitudes and values | Weeks 3 and 12
  Unvalidated questionnaires
Opinions about the study products | Weeks 6 and 12
  Unvalidated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marjukka Kolehmainen, Principal Investigator — University of Eastern Finland
Locations (1):
- Institute of Public Health and Clinical Nutrition, University of Eastern Finland, Kuopio, Finland